CLINICAL TRIAL: NCT03796715
Title: Comparison of Red Cell Distribution Width Versus Presepsin (Soluble CD14) for Prognosis Assessment in Sepsis Patients Admitted to the Intensive Care Unit
Brief Title: Red Cell Distribution Width Versus Presepsin (Soluble CD14) as a Prognostic Marker in Critically-ill Sepsis Patients
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed, Principal Investigator, Ain Shams University
Other Study IDs: FMASU R76/2018
Record Dates: First submitted 2019-01-01; First posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Sepsis
Keywords: sepsis; presepsin; red cell distribution width
MeSH Terms: conditions — Sepsis | interventions — Erythrocyte Indices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Red Cell Distribution Width (RDW): RDW was assessed as part of complete blood count analysis using SYSMEX XN-550 automated analyzer
  Interventions: Diagnostic Test: Red Cell Distribution Width (RDW)
- Presepsin (sCD14-ST): Presepsin analysis was done by utilising Elisa technique using kits from (MyBioSource, San Diego, CA 92195-3308 USA)
  Interventions: Diagnostic Test: Presepsin (sCD14-ST)

INTERVENTIONS:
Diagnostic Test: Red Cell Distribution Width (RDW) — A total of 100 sepsis patients, Red Cell Distribution Width (RDW) was used as prognostic marker.
  Groups: Red Cell Distribution Width (RDW)
Diagnostic Test: Presepsin (sCD14-ST) — : A total of 100 sepsis patients, Presepsin (sCD14-ST) was used as prognostic marker.
  Groups: Presepsin (sCD14-ST)

SUMMARY:
Presepsin (soluble CD14 subtype) is a novel marker with growing body of evidence supporting its accuracy and value for the diagnosis of sepsis. Patients with sepsis showed higher Prsepsin levels compared to those with SIRS. In addition the increase in Prsepsin levels correlates well with sepsis severity. Red cell distribution width variations are increased in a variety of medical conditions such as congestive heart failure, acute myocardial infarction, pulmonary embolism, pneumonia, critical illness, and cardiac arrest , and is a predictor of mortality in the general population. we aim to compare between Presepsin (soluble CD14) and RDW as prognostic markers in critically-ill patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 65 years.
* Appropriate clinical data to enable classification into sepsis or SIRS according to Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3).
* Written informed consent by the patient or guardian

Exclusion Criteria:

* No informed consent
* Renal failure
* Liver failure
* Hematologic diseases
* Neutropenia
* Malignancy
* Chemotherapy during the previous 90 days.
* Patients using antibiotics at presentation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the general ICU with sepsis or septic shock of both sexes between 18 and 65 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
Mortality during intensive care unit stay | 28 days

SECONDARY OUTCOMES:
Length of ICU stay | assessed up to 3 months
Need for readmission to ICU | assessed up to 3 months
Ventilatory support duration | assessed up to 3 months
Number of participants who need renal replacement therapy | assessed up to 3 months
Number of participants who need inotropic or vasopressor support | assessed up to 3 months
Transfusion requirements (blood and blood products) | assessed up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elsayed, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided